CLINICAL TRIAL: NCT04589806
Title: Evaluation of Bone Width Change Using a Two-stage Ridge Splitting Approach in Narrow Posterior Mandibular Ridge (Clinical Trial)
Brief Title: Change in Mandibular Bone Width Using Two Stages Splitting Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Narrow mandibular ridge
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Narrow Mandibular Ridge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-stage ridge splitting with simultaneous implant placement (Experimental)
  Interventions: Procedure: 2-stage ridge splitting

INTERVENTIONS:
Procedure: 2-stage ridge splitting — two-stage alveolar ridge splitting technique using piezoelectric device with simultaneous implant placement in order to treat narrow posterior mandibular ridges avoiding the risks of malfracture and necrosis of the split part

SUMMARY:
Alveolar ridge splitting technique is a commonly used procedure for horizontal ridge augmentation of narrow ridges to allow placement of implants. However, the commonly used one-stage technique can cause malfracture and subsequent necrosis of the fractured part.

DETAILED DESCRIPTION:
Twelve patients were selected randomly having posterior mandibular narrow edentulous ridge. The sample were selected to match a list of inclusion and exclusion criteria. In the first stage, all patients will underwent a mandibular ridge splitting technique using piezotomes. In the second stage, ridge expansion and implants were placed with only envelope flap. Assessment were included measurement of the buccal and lingual bone surrounding the implants and amount of increase in the bone width from the cone beam computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-60 years old with no gender predilection.
* Patients presenting with posterior mandibular (premolar-molar area) narrow alveolar ridge
* that requires dental implantation.
* Minimum bone width of 3 mm
* Minimum bone height of 10 mm
* Proper inter-occlusal space

Exclusion Criteria:

* Uncontrolled diabetes.
* Heavy smokers.
* Current chemotherapy or radiotherapy.
* Alcohol or drug abuse.
* Pregnant women.
* Active infection.
* Inter-occlusal space not less than 7-8 mm.
* Parafunctional habits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
change in the width of the alveolar bone | at the 1st week and the 4th month
  using CBCT the width were measured
Bone density | at the 4th week
  using CBCT the bone width were measured

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Eid, BDS, Principal Investigator — Researcher
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt